CLINICAL TRIAL: NCT05032443
Title: Awareness of Endoscopy Nurses Working in Pediatric Gastrointestinal Endoscopy Unit on Anesthesia Management; A Questionnaire Survey
Brief Title: Anesthesia Awareness in Pediatric Gastrointestinal Endoscopy Nurses
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Fatma Kartal, Responsible nurse, Ankara City Hospital Bilkent
Other Study IDs: E2-21-472
Record Dates: First submitted 2021-08-17; First posted 2021-09-02 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Endoscopy; Knowledge; Attitudes, Staff; Nurse's Role; Awareness, Anesthesia
Keywords: Pediatric endoscopy nurse; Awareness, Anesthesia; Questionnaire Survey
MeSH Terms: conditions — Behavior; Intraoperative Awareness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Awareness survey — The 33-item questionnaire will sent to pediatric endoscopy nurses in our country. Questionnaires will be delivered to nurses through hospital visits or electronic media.

SUMMARY:
Background and Aim: Pediatric gastrointestinal (GI) endoscopy is an increasingly common procedure performed to investigate and diagnose problems in the GI tract in children. Procedures in pediatric endoscopy units are routinely performed under sedation and general anesthesia, unlike adult endoscopy. Nurses working in pediatric gastroenoscopy units where sedoanalgesia is applied have important duties and responsibilities in terms of quality standards in preoperative, intraoperative and postoperative periods. Considering the increasing need for high-quality pediatric endoscopy applications, the attitudes and behaviors of nurses about sedation in pediatric patients are important as a member of the team. There is almost no literature on the experience and awareness of pediatric endoscopy nurses in clinical practice, and this encourages our team to conduct a survey across our country and to develop knowledge and clinical practices. With this questionnaire survey, it was aimed to evaluate the experience and attitudes of the endoscopy nurses working in the pediatric endoscopy unit in our country on sedation/general anesthesia management for pediatric patients

DETAILED DESCRIPTION:
Design: This research is a questionnaire survey. There will be no scaling in survey questions. The volunteers who will participate in the survey are nurses working in the pediatric endoscopy unit throughout Turkey, and the sample size was not calculated because it was desired to study in the whole universe and sampling was not used. Approximately 80 endoscopy nurses work in the pediatric endoscopy unit in Turkey. The universe consists of about 80 volunteers. Power analysis of the research will be done after the study is completed.

Methods: For this study, pediatric endoscopy nurses working in different clinics across our country will be invited. Questionnaires will be delivered to nurses through hospital visits or electronic media. The prepared questionnaire consists of a total of 33 questions evaluating nursing services on demographic data and sedation practices in pediatric endoscopy nurses' units. Of the 33 questions, 7 of them question the information about the socio-demographic data and professional experience of the pediatric endoscopy nurses, 16 of which will be answered as "yes" or "no" about the nursing services and approaches related to anesthesia management, the remaining 10 will consist of questions to be answered as "I agree" "I am undecided" "I do not agree".

ELIGIBILITY:
Inclusion Criteria:

* All pediatric endoscopy nurses working in the pediatric endoscopy unit in our country

Exclusion Criteria:

* Pediatric endoscopy nurses who will not want to participate in this questionnaire survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The volunteers who will participate in this questionnaire survey are nurses working in the pediatric endoscopy unit throughout Turkey
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Awareness survey | 30 minutes
  Evaluation of all pediatric endoscopy nurses' knowledge, awareness and attitudes about anesthesia management working in our country

SECONDARY OUTCOMES:
Developing a guideline | 30 minutes
  With this questionnaire study, it is desired to develop a guideline for the responsibility and awareness that should be created about anesthesia management in the clinic where pediatric endoscopy nurses work.
  The investigators would like to question the level of knowledge and awareness of the endoscopy nurse about anesthesia management in diagnostic and therapeutic procedures under sedation in the pediatric endoscopy unit and to organize training on the subjects that are deficient.
  Thus, the investigators aim to standardize quality pediatric endoscopy practices in every clinic in our country.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Kartal, Principal Investigator — Ankara City Hospital Bilkent; Feyza Sever, Study Director — Ankara City Hospital Bilkent; Şamil Hızlı, Study Director — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Çankaya, Turkey (Türkiye)